CLINICAL TRIAL: NCT01007331
Title: Probiotic Bacteria to Infants With Atopic Dermatitis; an Investigation of the Effect on Eczema, Immunologic Status and the Intestinal Microflora, Inflammation and Permeability
Brief Title: Probiotic Bacteria to Infants With Atopic Dermatitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Responsible Party: Kim Fleischer Michaelsen, Department of Human Nutrition, University of Copenhagen
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: KF-D200 Probørn
Record Dates: First submitted 2009-11-03; First posted 2009-11-04 (Estimated); Last update posted 2010-02-17 (Estimated); Status verified 2009-11

CONDITIONS: Atopic Dermatitis
Keywords: Infants; Atopic Dermatitis; SCORAD; IgE; Eosinophil Cation Protein; Calprotectin; Intestinal microflora
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Lactobacillus acidophilus NCFM and Bifidobacterium lactis Bi-07 — 10^10 colony forming units pr day of probiotics

SUMMARY:
The objective of the study is to examine whether 8 weeks intervention with probiotics influence the eczema in infants suffering from Atopic Dermatitis. Furthermore the influence of the immunologic status and the intestinal microflora, inflammation and permeability will be investigated.

DETAILED DESCRIPTION:
The aim of the study is to investigate whether two different probiotics influence the clinical and subjective symptoms in infants with Atopic Dermatitis (AD). The influence on the immunologic status and the intestinal microflora, inflammation and permeability will also be investigated.

Sixty two infants (6 to 24 months of age) suffering from AD will be randomised in 3 groups receiving either Lactobacillus acidophilus NCFM (1x10^10 Colony forming units), Bifidobacterium lactis Bi-07(1x10^10 Colony forming units) or placebo every day for 8 weeks.

At the beginning and at the end of the study the following analyses will be made:

1. SCORing Atopic Dermatitis (SCORAD) index to describe the extent and severity of the eczema, and to describe the subjective symptoms.
2. Blood samples will be drawn to examine:

   * Immunoglobulin E (IgE), total and specific for egg and milk.
   * Eosinophil Cation Protein (ECP)
   * Interleukin-10 (Il-10), Interleukin-12 (Il-12) and Interferon-gamma (IFN-gamma)
3. Fecal samples will be collected to examine:

   * Calprotectin (intestinal inflammation)
   * Bacterial Deoxyribonucleic acid (DNA) will be extracted in order to perform Polymerase chain reaction (PCR) analysis.

ELIGIBILITY:
Inclusion Criteria:

* Atopic dermatitis

Exclusion Criteria:

* Chronic diseases other than atopic dermatitis
* Chronic medication

Ages: 6 Months to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 62 (Actual)
Dates: Start 2006-11; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Scoring atopic dermatitis (SCORAD) index | 5 months

SECONDARY OUTCOMES:
Immunoglobulin E (IgE) Total | 6 months
Immunoglobulin E (IgE) specific for Egg | 6 months
Immunoglobulin E (IgE) specific for Milk | 6 months
Interleukin-10 (Il-10) | 6 months
Interleukin-12 (Il-12) | 6 months
Interferon gamma (IFN-gamma) | 6 months
Calprotectin | one year
Polymerase Chain Reaction (PCR) | 8 months
Eosinophil Cation Protein (ECP) | 7 months

CONTACTS AND LOCATIONS:
Overall Officials: Kim F Michaelsen, Professor, Principal Investigator — Department of Human Nutrition, University of Copenhagen
Locations (1):
- Institute of Human Nutrition, Rolighedsvej 30, Frederiksberg C, Denmark